CLINICAL TRIAL: NCT06844786
Title: SCORE! ACTIVE: Advancing Codesigned Health Promotion and Physical Activity Interventions to Improve Self-Efficacy and Health: A Stepped Wedge Cluster Randomized Trial
Brief Title: SCORE! ACTIVE Trial
Acronym: ACTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Gita Wahi, Associate Professor, Pediatrics, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17739
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Disease; Childhood Obesity
MeSH Terms: conditions — Chronic Disease; Pediatric Obesity | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCORE! ACTIVE (Experimental): This is the only arm of the study. The interventions included in this arm are physical activity programming (SCORE! CLUB), navigator services (SCORE! navigator), and health promotion messaging. All clusters will receive this intervention.
  Interventions: Other: Physical activity program; Other: Navigation; Other: Health promotion

INTERVENTIONS:
Other: Physical activity program — SCORE! Club is offered twice a week for enrolled participants. Modules will include soccer, arts and health, Sportball, and nature-based activities.
  Other Names: SCORE! Club
Other: Navigation — Participants will have access to a navigator from the study team who will help them access resources relating to recreation and physical activity in their communities. For example, the navigator will help direct families with low income to the recreation assistance program if they are interested in such a service.
  Other Names: SCORE! Navigator
Other: Health promotion — Health promotion messaging will be provided to participants via social media and other physical methods (i.e., flyers). Topics will include diet, sleep, physical activity, and other related items.
  Other Names: Health promotion messaging

SUMMARY:
Hamilton is a city with a growing newcomer population. Families who are new to Canada do not always have the same resources to access healthy active living (HAL) activities as compared to Canadian-born families. The SCORE! ACTIVE trial will recruit newcomer families with young children in Hamilton and help provide them with access to HAL activities. Through this, the investigators want to see if newcomer children's perspectives of physical activity will change over time. They will also see if increasing newcomer children's access to these resources will promote an increase in HAL behaviours.

DETAILED DESCRIPTION:
The investigators will conduct a pragmatic, stepped-wedge cluster randomized trial in 14 neighbourhoods to determine the impact of SCORE! ACTIVE trial on the primary outcome of PA self-efficacy among 5-11-year-old children. The SW-CRT involves the sequential transition of clusters, in this case neighbourhoods, from control to intervention conditions in a randomized order. In this case, the method is pragmatic because recruitment and initial baseline measures in each community will occur just before the initiation of the intervention. There have been methodological challenges noted with SW-CRT including identification and recruitment bias, within cluster bias, and secular trends. However, this design is ideal for the implementation of the SCORE! ACTIVE trial because for practical reasons, it is not possible to deliver the intervention to many clusters at the same time. The trial will be reported using CONSORT guidelines and extension of SW-CRT.

ELIGIBILITY:
Inclusion Criteria:

* Newcomer families (those who have been in Canada for 10 years or less) with at least 1 child aged 5 up to 11 (11.99 years) living in a Hamilton, Ontario.
* At least one parent/guardian born outside of Canada and residing in Canada ≤ 10 years.
* Families must be living in one of the designated neighbourhood clusters

Exclusion Criteria:

* Children participating in organized physical activity programs for 3 or more times per week
* Families with involvement with child protection services and/or foster care

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1400 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Children's Self-Perceptions of Adequacy in and Predilection for Physical Activity (CSAPPA) Scale | Baseline to 6 months
  Using CSAPPA, a 19-item scale that measures how children feel about their physical activity skills and their likelihood of choosing physical activities, a change in children's physical activity self-efficacy will be measured at 6 months as the primary outcome.

SECONDARY OUTCOMES:
Children's Self-Perceptions of Adequacy in and Predilection for Physical Activity (CSAPPA) Scale | 12 months from baseline; 18 months from baseline
  Using CSAPPA, a change in children's physical activity self-efficacy will also be measured at 12 and 18 months as secondary outcomes.
Physical Activity & Sedentary Behavior Questionnaire | Baseline to 18 months
  Changes in children's physical activity and sedentary behaviours will be measured using the Physical Activity & Sedentary Behavior Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No